CLINICAL TRIAL: NCT01361828
Title: Electrophysiological Assessment of Optic Nerve and Retinal Functions Following Intravitreal Injection of Bevacizumab (Avastin).
Brief Title: Optic Nerve and Retinal Functions With Bevacizumab
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Tamer A Macky, Cario University
Other Study IDs: Beva-ERG-VEP
Record Dates: First submitted 2011-05-26; First posted 2011-05-27 (Estimated); Last update posted 2011-05-27 (Estimated); Status verified 2010-01

CONDITIONS: Choroidal Neovascular Membrane
Keywords: Bevacizumab; VEP; ERG; Optic nerve and retinal functions following intravitreal bevacizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with choroidal neovascularization: CNV due to Age-Related Macular Degenerations and Myopia were included.
  Interventions: Procedure: Electrophysiology

INTERVENTIONS:
Procedure: Electrophysiology — Visual Evoked Potential and Elctroretinogram

SUMMARY:
The purpose of this study is to investigate the possible affection of optic nerve and retinal functions following intravitreal bevacizumab injection in human eyes.

DETAILED DESCRIPTION:
To evaluate the retinal and optic nerve functions of bevacizumab when injected intravitreal in human eyes using electrophysiological tests; Electroretinogram (ERG) and Visual Evoked Potentials (VEP). Forty five eyes of 45 patients with choroidal neovascular membrane (CNV) who were prepared for intravitreal injections of 1.25mg bevacizumab underwent baseline ERG and VEP in both eyes before, and at 1 and 4 weeks after the intravitreal injections.

ELIGIBILITY:
Inclusion Criteria:

* CNV

Exclusion Criteria:

* Previous Intravitreal Injections

Ages: 24 Years to 62 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Forty five eyes of 45 patients with choroidal neovascular membrane (CNV) who were prepared for intravitreal injections of 1.25mg bevacizumab underwent baseline ERG and VEP in both eyes before, and at 1 and 4 weeks after the intravitreal injections.Mean age was 50 years ranging from 24-62 years with 25 females, with 28 AMD and 17 myopic patients.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2010-01; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Visual Evoked Potential and Electroretinogram | 4 weeks
  VEP and ERG baseline and at 1 and 4 weeks post intravitreal injection of bevacizumab.

CONTACTS AND LOCATIONS:
Overall Officials: Tamer A macky, Principal Investigator — Cairo University
Locations (1):
- Cairo University, Cairo, --- Select One ---, Egypt

REFERENCES:
- See also: Electrophysiological assessment of retinal function during 6 months of bevacizumab treatment in neovascular age-related macular degeneration. — http://www.ncbi.nlm.nih.gov/pubmed/20616681